CLINICAL TRIAL: NCT03936127
Title: Comparison of a Novel Transperineal Targeted Fusion Biopsy System to Conventional Transrectal Targeted Fusion Biopsy for Diagnosis of Clinically Significant Prostate Cancers and to Eliminate Post-procedure Related Infections: A Randomized Control Trial
Brief Title: Comparison of a Novel Transperineal Targeted Fusion Biopsy System to Conventional Transrectal Targeted Fusion Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Nicola Schieda (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor-Investigator, Dr. Nicola Schieda, Director of Abdominal and Pelvic MRI, The Ottawa Hospital, The Ottawa Hospital
Organization: The Ottawa Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20190262-01H
Record Dates: First submitted 2019-04-25; First posted 2019-05-03 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: Transperineal; Transrectal; Fusion Biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperineal (TP) Ultrasound (US) Targeted Fusion Biopsy (Experimental): Transperineal (TP) ultrasound (US) targeted fusion biopsy (which is performed using a validated Health Canada approved elastic software fusion platform).
  Interventions: Procedure: Ultrasound (US) Targeted Fusion Biopsy
- Transrectal (TR) Ultrasound (US) Targeted Fusion Biopsies (Active Comparator): Transrectal (TR) ultrasound (US) targeted fusion biopsy (which is performed using a validated Health Canada approved elastic software fusion platform).
  Interventions: Procedure: Ultrasound (US) Targeted Fusion Biopsy

INTERVENTIONS:
Procedure: Ultrasound (US) Targeted Fusion Biopsy — Ultrasound (US) Targeted Fusion Biopsy

SUMMARY:
This study is designed as a randomized control trial which intends to determine if transperineal (TP) targeted biopsy is not inferior to transrectal (TR) targeted biopsy for diagnosis of clinically significant prostate cancer while comparing post-procedural infection rates between the two techniques. The study will also look to compare patient reported pain scores related to the procedure, rates of other minor complications (e.g. bleeding, urinary retention) and procedure time.

The expected sample size at The Ottawa Hospital is 360 men.

DETAILED DESCRIPTION:
Patients undergo mp-MRI, at the discretion of the treating Urologist, when they are referred to the Cancer Assessment Clinic for their initial visit with a risk factor for prostate cancer (e.g. abnormal digital rectal exam [DRE] or elevated prostate serum antigen [PSA] level). Performing an mp-MRI in a man with risk factors for prostate cancer prior to an initial biopsy has become the standard of care for diagnosis of prostate cancer based on two large multi-center randomized control trials.

At the second visit, which is standard of care, the Urologist (or delegate [Resident, Fellow]) will discuss targeted biopsy and will introduce the trial design obtaining informed consent to participate. If consent is obtained, the patient will be randomly assigned to receive either the standard transrectal (TR) ultrasound guided targeted fusion biopsy or the novel transperineal (TP) targeted fusion biopsy system which has also been preliminarily validated as being accurate for detection of significant prostate cancers at targeted biopsy.

Patients will be notified regarding which method of targeted biopsy will be employed at time of scheduling.

Both the TR and TP biopsies will be conducted in existing biopsy rooms in The Ottawa Hospital (TOH) and will employ a brief 30-minute post-procedural observation period at which point the patient is required to urinate prior to discharge. Level of pain will be recorded by the ultrasound technologists during the 30 minutes observation period as well.

This study aims to compare ultrasound guided transrectal and transperineal targeted fusion biopsy for diagnosis of prostate cancer in abnormalities detected on MRI for the purpose of reducing or completely eliminating the risk of serious infection associated with the transrectal approach.

ELIGIBILITY:
Inclusion Criteria:

* MRI positive - abnormal area detected
* Patient re-evaluated in the TOH Prostate CAC (Cancer Assessment Centre) for planning of targeted biopsy
* Signed Consent

Exclusion Criteria:

* MRI negative - no abnormal area detected
* Patient with a prior diagnosis of prostate cancer enrolled in active surveillance

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The expected sample size at The Ottawa Hospital is 360 men.
Enrollment: 360 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Infection Rate | Patients who have undergone biopsy of the prostate will be seen by their Urologist in routine clinical follow-up, typically in 4-6 weeks, as per standard of care.
  Number of patients with or without post-procedural infection.

SECONDARY OUTCOMES:
Clinically Significant Prostate Cancer | Patients who have undergone biopsy of the prostate will be seen by their Urologist in routine clinical follow-up, typically in 4-6 weeks, as per standard of care.
  Gleason score of tumor in biopsy samples containing cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Schieda, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Time Frame: The Principal Investigator will aim to have data available within 12 months of study completion.
Access Criteria: * Authors aim to have the study presented at conferences and published in a peer-reviewed journal.
  * Authors aim to have the study presented at conferences and published in a peer-reviewed journal.
  * A description of this clinical trial/study will be available on http://www.clinicaltrials.gov. Participants can search this website at anytime to obtain all study information.
URL: http://www.clinicaltrials.gov.

REFERENCES:
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Nam RK, Saskin R, Lee Y, Liu Y, Law C, Klotz LH, Loblaw DA, Trachtenberg J, Stanimirovic A, Simor AE, Seth A, Urbach DR, Narod SA. Increasing hospital admission rates for urological complications after transrectal ultrasound guided prostate biopsy. J Urol. 2013 Jan;189(1 Suppl):S12-7; discussion S17-8. doi: 10.1016/j.juro.2012.11.015. PMID 23234616
- [Background] Rudzinski JK, Kawakami J. Incidence of infectious complications following transrectal ultrasound-guided prostate biopsy in Calgary, Alberta, Canada: A retrospective population-based analysis. Can Urol Assoc J. 2014 May;8(5-6):E301-5. doi: 10.5489/cuaj.1751. PMID 24940454
- [Background] Guo LH, Wu R, Xu HX, Xu JM, Wu J, Wang S, Bo XW, Liu BJ. Comparison between Ultrasound Guided Transperineal and Transrectal Prostate Biopsy: A Prospective, Randomized, and Controlled Trial. Sci Rep. 2015 Nov 3;5:16089. doi: 10.1038/srep16089. PMID 26526558
- [Background] Verma S, Choyke PL, Eberhardt SC, Oto A, Tempany CM, Turkbey B, Rosenkrantz AB. The Current State of MR Imaging-targeted Biopsy Techniques for Detection of Prostate Cancer. Radiology. 2017 Nov;285(2):343-356. doi: 10.1148/radiol.2017161684. PMID 29045233
- [Background] Barrett T, Haider MA. The Emerging Role of MRI in Prostate Cancer Active Surveillance and Ongoing Challenges. AJR Am J Roentgenol. 2017 Jan;208(1):131-139. doi: 10.2214/AJR.16.16355. Epub 2016 Oct 11. PMID 27726415
- [Background] Kosarek CD, Mahmoud AM, Eyzaguirre EJ, Shan Y, Walser EM, Horn GL, Williams SB. Initial series of magnetic resonance imaging (MRI)-fusion targeted prostate biopsy using the first transperineal targeted platform available in the USA. BJU Int. 2018 Nov;122(5):909-912. doi: 10.1111/bju.14206. Epub 2018 Apr 14. PMID 29569311
- [Background] Costa DN, Kay FU, Pedrosa I, Kolski L, Lotan Y, Roehrborn CG, Hornberger B, Xi Y, Francis F, Rofsky NM. An initial negative round of targeted biopsies in men with highly suspicious multiparametric magnetic resonance findings does not exclude clinically significant prostate cancer-Preliminary experience. Urol Oncol. 2017 Apr;35(4):149.e15-149.e21. doi: 10.1016/j.urolonc.2016.11.006. Epub 2016 Dec 9. PMID 27939349
- [Background] Oderda M, Faletti R, Battisti G, Dalmasso E, Falcone M, Marra G, Palazzetti A, Zitella A, Bergamasco L, Gandini G, Gontero P. Prostate Cancer Detection Rate with Koelis Fusion Biopsies versus Cognitive Biopsies: A Comparative Study. Urol Int. 2016;97(2):230-7. doi: 10.1159/000445524. Epub 2016 Jun 4. PMID 27256369
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Schmit GD, Schenck LA, Thompson RH, Boorjian SA, Kurup AN, Weisbrod AJ, Kor DJ, Callstrom MR, Atwell TD, Carter RE. Predicting renal cryoablation complications: new risk score based on tumor size and location and patient history. Radiology. 2014 Sep;272(3):903-10. doi: 10.1148/radiol.14132548. Epub 2014 May 7. PMID 24814178
- See also: Canadian Cancer Society (2018) Canadian Cancer Statistics — http://www.cancer.ca/en/cancer-information/cancer-type/prostate/statistics/?region=on